CLINICAL TRIAL: NCT00299832
Title: A Multi-center, Open-label Study Assessing the Safety, Efficacy and Pharmacokinetics of 8 Week's Treatment of SPP100 (Aliskiren) Regimen in Hypertensive Patients With Renal Dysfunction
Brief Title: SPP100 (Aliskiren) Regimen in Hypertensive Patients With Renal Dysfunction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100A1303
Record Dates: First submitted 2006-03-03; First posted 2006-03-07 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, blood pressure, rennin
MeSH Terms: conditions — Hypertension | interventions — aliskiren

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Aliskiren

SUMMARY:
Assessing the safety, efficacy and pharmacokinetics of SPP100 (Aliskiren) regimen in hypertensive patients with renal dysfunction

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 - 80 years old
* Gender: Male or female
* Status: Outpatients
* Elevated Serum Creatinine

Exclusion Criteria:

* Patients suspected of malignant hypertension
* Patients with a clinically significant allergy
* Patients who have received other investigational drug Other protocol-defined inclusion/exclusion criteria may apply

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Adverse events after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure after 8 weeks
Change from baseline in mean sitting diastolic blood pressure after 8 weeks
Mean sitting systolic blood pressure is < 140 mmHg or a reduction of > 20 mmHg after 8 weeks
Mean sitting diastolic blood pressure is < 90 mmHg or a reduction of > 10 mmHg after 8 weeks
Blood pressure <140/90 after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Novartis Pharmaceuticals, Japan, Japan

REFERENCES:
- [Result] Ito S, Nakura N, Le Breton S, Keefe D. Efficacy and safety of aliskiren in Japanese hypertensive patients with renal dysfunction. Hypertens Res. 2010 Jan;33(1):62-6. doi: 10.1038/hr.2009.175. Epub 2009 Nov 20. PMID 19927154